CLINICAL TRIAL: NCT06257459
Title: Excision Versus Preservation of Spermatic Cord Lipoma Detected During Subinguinal Varicocelectomy in Infertile Men With Oligo-asthenzoospermia: A Prospective Randomized Trial.
Brief Title: Excision Versus Preservation of Spermatic Cord Lipoma Detected During Subinguinal Varicocelectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Zoeir, faculty of medicine, Tanta, ElGeish street, Egypt, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 36137/12/22
Record Dates: First submitted 2024-01-30; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Male Infertility
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lipoma Excision (group A) (Active Comparator): excison of spermatic cord lipoma detected during subinguinal varicocelectomy in infertile males
  Interventions: Procedure: subinguinal varicocelectomy
- Lipoma Preservation (group B) (Active Comparator): preservation of spermatic cord lipoma detected during subinguinal varicocelectomy in infertile males
  Interventions: Procedure: subinguinal varicocelectomy

INTERVENTIONS:
Procedure: subinguinal varicocelectomy — exision or preservation of spermatic cord lipoma during subinguinal varicocelectomy

SUMMARY:
In the current study, the adult infertile patients with clinical varicoceles will be included. the patients will undergo subinguinal varicocelectomy. The patients with spermatic cord lipoma detected at the time of surgery will be enrolled and divided into 2 groups( excision group, group A and preservation group (B). semen parameters will be compared in both group at 3 and 6 months after surgery

DETAILED DESCRIPTION:
This will be a prospective randomized study, in which adult infertile patients with clinical varicocele and oligo-athenospermia admitted to Urology department Tanta university hospital will be included and then the patients with detected spermatic cord lipoma at the time surgery will be enrolled and divided into 2 groups:

GROUP A : will undergo subinguinal varicocelectomy with excision of spermatic cord lipoma GROUP B : will undergo subinguinal varicocelectomy with preservation of spermatic cord lipoma

Inclusion criteria:

* Adult infertile males
* Clinical varicocele
* oligo-asthenospermia

Exclusion criteria:

* Adolescent varicocele
* Recurrent varicocele
* Presence of inguinal hernia
* Azospermic patients

ELIGIBILITY:
Inclusion Criteria:

* Adult infertile males
* Clinical varicocele
* Semen analysis show oligo-athenospermia

Exclusion Criteria:

* Adolescent varicocele
* Recurrent varicocele
* Presence of inguinal hernia
* Azospermic patients

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
semen parameters improvement | 3 and 6 months after surgery
  semen analysis
symptoms improvement (pain and swelling) | 3 and 6 months after surgery
  improvement of preoperative scrotal pain and swelling was assessed

SECONDARY OUTCOMES:
postoperative complications | early after surgery and late
  post-operative scrotal edema, hematoma and wound infection were assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Zoeir, Tanta, Gharbia Governorate, Egypt